CLINICAL TRIAL: NCT05389202
Title: Study of Prostate Perfusion Before Embolization in Patients With Symptomatic Prostate Adenoma. A Single-center Prospective Cohort Pilot Study to Determine the Predictive Factors of Clinical Efficacy Associated With a Prior Phantom Study.
Brief Title: Study of Prostate Perfusion Before Embolization in Patients With Symptomatic Prostate Adenoma
Acronym: EMBOPERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2021-1/JF-01
Record Dates: First submitted 2022-05-11; First posted 2022-05-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Prostate; Adenoma; Embolization
MeSH Terms: conditions — Prostatic Neoplasms; Adenoma

STUDY DESIGN:
Masking Description: The infusion scans will be interpreted by a radiologist who does not know the patient's clinical result in order to avoid a classification bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients benefitting from a perfusion CT scan before embolization (Experimental): Prostatic perfusion parameters seem to be correlated with the effectiveness of embolization. Studying these prostatic perfusion parameters in perfusion CT and evaluating the prostatic Iodine load in dual energy CT will make it possible to better select responder patients.
  Interventions: Other: Perfusion CT scanning

INTERVENTIONS:
Other: Perfusion CT scanning — Abdominopelvic CT scan with perfusion and spectral analysis performed 7 days (± 5 days) before prostate embolization.

SUMMARY:
Over the last 5 years, prostate embolization has developed as a treatment for symptomatic prostate adenoma. This long, complex procedure is effective in 80% of cases. Currently there are no means of better selecting patients to avoid this long procedure in non-responders. The hypothesis is that prostate perfusion parameters are correlated with the efficacy of embolization. Studying these prostate perfusion parameters in perfusion CT and evaluating prostate Iodine load in dual energy computed tomography will make it easier to select those patients who are most likely to respond.

DETAILED DESCRIPTION:
The hypothesis is that there are two types of prostate vascularization in patients with symptomatic prostate adenoma:

* prostates mainly vascularized by large caliber prostate arteries with high flow, for which perfusion parameters in favor of hyper-perfusion will be found. In this case, prostate artery embolization will be effective;
* prostates vascularized by a network of collaterals, with low flow-rates, for which perfusion parameters in favor of hypo-perfusion will be found. In this case, prostate artery embolization will not be very effective.

The purpose of this study is to investigate the association between prostate perfusion parameters (peak time, transit time, blood volume, capillary permeability) and the clinical efficacy of prostate embolization at 3 months. These perfusion parameters could become new biomarkers leading to better selection of patients eligible for efficient prostate embolization, in order to avoid a considerable treatment with no benefit for certain patients and thus limit their global exposure to X-rays during care.

Prior to this prospective study on patients with symptomatic benign prostate hypertrophy, a preliminary experimental study will be performed on a perfusion phantom in order to better understand the differences in the calculation of perfusion parameters according to the three main algorithms used. This will lead to optimization of the prostate perfusion protocol for the scanner: computed tomography acquisition parameters (kilovoltage, Milliamps per second) and therefore the X-ray dose delivered to patients, sampling frequency, and model to be used. The first results of this study have already led to modifications in scanner perfusion acquisition protocols for the initiation of clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic benign prostatic hypertrophy (prostate volume > 50, IPSS >7, QoL>2) or patients catheterized after acute retention of urine with failed catheterization.
* Creatinine clearance > 30 mL/min for one of the two Cockcroft-Gault/MDRD equations)
* Adult patients (≥18 years).
* Patients with an indication for prostate embolization.
* Patient with free and informed consent.
* Patient who have signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* Hypersensitivity to the active substance or to one of the excipients of the iodized contrast medium.
* Severe renal impairment with renal function <30mL/min.
* Contraindication to prostate embolization (aorto-iliac bypass)
* Patient participating in research defined as Category 1 Research Involving Human Subjects.
* Patient in an exclusion period as determined by another study.
* Patient under court protection, guardianship or curatorship.
* Patient unable to give consent.
* Patient for whom it is impossible to give informed information.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males only
Enrollment: 45 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Catheterized patients: Removal of the urinary catheter at 3 months | Month 3
  Yes/No
Non-catheterized patients: 25% decrease in the International Prostate Symptom Score | Month 3
  Yes/No
Non-catheterized patients: one point improvement in the Global Quality of Life Score. | Month 3
  Yes/No
MRI perfusion parameters : Capillary permeability | 7 - 14 days before embolization
  Measured in mL.mL tissue-1.min-1
Scanner perfusion parameters : Capillary permeability | Day 0 (on the day of embolization)
  Measured in mL.mL tissue-1.min-1
MRI perfusion parameters : Extracellular volume | 7 - 14 days before embolization
  Measured in mL.mL tissue-1
Scanner perfusion parameters : Extracellular volume | Day 0 (on the day of embolization)
  Measured in mL.mL tissue-1
MRI perfusion parameters : Blood volume | 7 - 14 days before embolization
  Measured in mL.mL tissue-1
Scanner perfusion parameters : Blood volume | Day 0 (on the day of embolization)
  Measured in mL.mL tissue-1
MRI perfusion parameters : Maximum slope | 7 - 14 days before embolization
  Measured in ml.min-1
Scanner perfusion parameters : Maximum slope | Day 0 (on the day of embolization)
  Measured in ml.min-1
MRI perfusion parameters : Time to peak | 7 - 14 days before embolization
  Measured in seconds
MRI perfusion parameters : Time to peak | Day 0 (on the day of embolization)
  Measured in seconds
Scanner perfusion parameters : Prostate iodine load at 80 s. | 7 - 14 days before embolization
  Measured in mgI.mg of prostate-1
MRI perfusion parameters : Prostate iodine load at 80 s. | Day 0 (on the day of embolization)
  Measured in mgI.mg of prostate-1

SECONDARY OUTCOMES:
Influence of flow rate on the scanner algorithm | 1 - 15 days before embolization. Preliminary stage on phantom.
  The influence of flow rate on the scanner algorithm will be measured on the perfusion phantom model in mL.min-1.
A. Correspondence between MRI and scanner: Capillary permeability | 1 - 7 days before embolization
  Measured in mL.mL tissue-1.min-1
A. Correspondence between MRI and scanner: Extracellular volume | 1 - 7 days before embolization
  Measured in mL.mL tissue-1
A. Correspondence between MRI and scanner: Blood volume | 1 - 7 days before embolization
  Measured in mL.mL tissue-1
A. Correspondence between MRI and scanner: Maximum slope | 1 - 7 days before embolization
  Measured in mL.min-1
A. Correspondence between MRI and scanner: Time to peak | 1 - 7 days before embolization
  Measured in seconds
A. Correspondence between MRI and scanner: 80-second iodine load | 1 - 7 days before embolization
  Measured in mgl.mg of prostate-1
B. 4-D map Magnetic Resonance Imaging perfusion parameters : Volume of beads injected | At the time of embolization
  Measured in mL
B. Scanner perfusion parameters : Volume of beads injected | At the time of embolization
  Measured in mL
C. Influence of scanner acquisition parameters: kV | 1 to 15 days before embolization. Preliminary stage on phantom.
  The influence of scanner acquisition parameters on the scanner algorithm will be measured on the the perfusion phantom model.
C. Influence of scanner acquisition parameters: mAs | 1 to 15 days before embolization. Preliminary stage on phantom.
  The influence of scanner acquisition parameters on the scanner algorithm will be measured on the the perfusion phantom model.
C. Influence of scanner acquisition parameters: iterative reconstruction | 1 to 15 days before embolization. Preliminary stage on phantom.
  The influence of scanner acquisition parameters on the scanner algorithm will be measured on the the perfusion phantom model.
C. Blood volume | 1 to 15 days before embolization. Preliminary stage on phantom.
  The perfusion parameter "blood volume" will be measured on the phantom in mL
C. Maximum slope | 1 to 15 days before embolization. Preliminary stage on phantom.
  The perfusion parameter "maximum slope" will be measured on the phantom in mL.min-1
C. Time to peak | 1 to 15 days before embolization. Preliminary stage on phantom.
  The perfusion parameter "time to peak" will be measured on the phantom in seconds

OTHER OUTCOMES:
Age | Day 0
  In years
Weight | Day 0
  In kilograms
Height | Day 0
  In centimeters
Comorbidities | Day 0
  All comorbidities such as cardiovascular condition, smoking etc., and diabetes will be recorded on the electronic patient file.
Adverse events | Day 0
  Any adverse events will be recorded: Allergy to contrast medium, urinary tract sepsis, persistent urinary tract infection, dysuria, severe hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectal bleeding, severe radiation skin injury, acute urinary retention, pelvic-perineal pain, acute urinary retention, prostatitis, orchi-epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder. Puncture site hematoma, artery dissection/vessel injury (dissection, perforation, rupture, occlusion, spasm), false aneurysm requiring intervention, arteriovenous fistula requiring intervention, angioplasty or stenting, hematoma/bleeding requiring transfusion or surgery, arterial embolism/thrombosis, need for revascularization by bypass surgery, infection. Due to dual-energy CT with contrast injection: stochastic risk of X-ray exposure; risks related to non-ionic contrast injection: intolerance, nausea, vomiting, urticaria, anaphylactic shock.
Adverse events | Day 7
  Any adverse events will be recorded: Allergy to contrast medium, urinary tract sepsis, persistent urinary tract infection, dysuria, severe hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectal bleeding, severe radiation skin injury, acute urinary retention, pelvic-perineal pain, acute urinary retention, prostatitis, orchi-epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder. Puncture site hematoma, artery dissection/vessel injury (dissection, perforation, rupture, occlusion, spasm), false aneurysm requiring intervention, arteriovenous fistula requiring intervention, angioplasty or stenting, hematoma/bleeding requiring transfusion or surgery, arterial embolism/thrombosis, need for revascularization by bypass surgery, infection. Due to dual-energy CT with contrast injection: stochastic risk of X-ray exposure; risks related to non-ionic contrast injection: intolerance, nausea, vomiting, urticaria, anaphylactic shock.
Adverse events | Month 3
  Any adverse events will be recorded: Allergy to contrast medium, urinary tract sepsis, persistent urinary tract infection, dysuria, severe hematuria, hemospermia, bladder ulceration/necrosis, rectal ulcer, rectal bleeding, severe radiation skin injury, acute urinary retention, pelvic-perineal pain, acute urinary retention, prostatitis, orchi-epididymitis, obstructive renal failure, chronic bladder retention, lithiasis, hypocontractile bladder. Puncture site hematoma, artery dissection/vessel injury (dissection, perforation, rupture, occlusion, spasm), false aneurysm requiring intervention, arteriovenous fistula requiring intervention, angioplasty or stenting, hematoma/bleeding requiring transfusion or surgery, arterial embolism/thrombosis, need for revascularization by bypass surgery, infection. Due to dual-energy CT with contrast injection: stochastic risk of X-ray exposure; risks related to non-ionic contrast injection: intolerance, nausea, vomiting, urticaria, anaphylactic shock.

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France